CLINICAL TRIAL: NCT02613702
Title: Efficacy of a Modified Technique of Free Gingival Graft in Volumetric Changes of the Graft: Randomized Clinical Trial
Acronym: EFFECT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Universidade Estadual de Maringá (Other)
Responsible Party: Principal Investigator, Claudio Mendes Pannuti, Associate Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFFECT
Record Dates: First submitted 2015-11-18; First posted 2015-11-24 (Estimated); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Gingival Recession
Keywords: Free gingival graft; keratinized gingival tissue
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Modified Free Gingival Graft (Experimental): Twenty patients will receive the modified free gingival graft technique at the inferior incisors area. In this technique, the graft is covered by a flap, similarly to what is done in a connective tissue graft surgery.
  Interventions: Procedure: Free Gingival Graft; Procedure: Modified Free Gingival Graft technique
- Original Free Gingival Graft technique (Active Comparator): Twenty patients will receive the original technique of free gingival graft at the inferior incisors area.
  Interventions: Procedure: Free Gingival Graft; Procedure: Original Free Gingival Graft technique

INTERVENTIONS:
Procedure: Free Gingival Graft — Surgical technique (autologous graft): Free gingival graft technique, harvested from palate.
Procedure: Original Free Gingival Graft technique — Surgical technique (autologous graft): Original technique of free gingival graft, positioned at the inferior incisors area at the donor area
  Arms: Original Free Gingival Graft technique
Procedure: Modified Free Gingival Graft technique — Surgical technique (autologous graft): Free gingival graft. positioned at the inferior incisors area and covered by a flap at the donor area
  Arms: Modified Free Gingival Graft

SUMMARY:
This study will compare a new technique of free gingival graft to the original one, in order to evaluate the stability of the graft volume over one year and other variables. Twenty patients will receive the original technique of free gingival graft (controls) and twenty patients will receive the modified technique, in which the free gingival graft is submerged (tests), at the inferior incisors area.

DETAILED DESCRIPTION:
The free gingival graft surgery is held to gain some keratinized tissue in areas where it has been lost, such as in inferior incisors with gingival recessions. In these areas, tooth brushing may become harder and painful, negatively influencing in plaque control. However, this type of graft seems to contract over time. A new approach of free gingival graft, in which the graft is covered by a flap, promises to provide greater vascularization. This would promote less graft contraction and better mucosal color. Forty patients with less than 2 mm of keratinized tissue (measured from gingival margin to mucogingival junction) in at least one inferior incisor will be included. Half will receive the original technique and half will receive the modified one. Patients will be followed at 7, 14, 21, 28, 42 days, 3, 6, 12 months and 8 years after surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Reduced keratinized tissue (less than 2 mm) in inferior incisors area
* Healthy periodontium in inferior incisors area
* Indication for surgery (e.g. pain during tooth brushing, gingival margin mobility, gingival recession...)
* Recessions class I, II or III, maximum 3 mm
* Having signed the informed consent

Exclusion Criteria:

* Systemic diseases
* Smokers
* Pregnant and lactating women
* Root caries lesions
* Previous surgeries at same area
* Accentuated root abrasion
* Malpositioning teeth
* Residual pocket depths greater than 4 mm
* Tooth mobility greater than 1

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-09 (Actual); Primary Completion 2025-05 (Actual); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Apical-cervical width of keratinized tissue after 12 months | 12 months
  Distance between gingival margin and mucogingival junction, in millimeters

SECONDARY OUTCOMES:
Probing Depth | 12 months
  Distance between gingival margin and bottom of the sulcus / pocket, in millimeters
Keratinized tissue area | 12 months
  Keratinized tissue area, measured in millimeters
Keratinized tissue thickness | 12 months
  Keratinized tissue thickness measured in millimeters
Volume of receiving area | 12 months
  Volume of receiving area
Complete epithelization of donor area | 28 days
  Area of Epithelization of wound healing, measured in mm2
Postoperative discomfort | 28 days
  discomfort measured using Visual Analogue Scale
Gum color | 12 months
  Measured with photographic analysis
Oral Health Related Quality of Life (OHIP) | 12 months
  OHIp - 14 short version
Clinical Attachment Level | 12 months
  Distance between cementum-enamel junction and bottom of sulcus / pocket, measured in millimeters
Recession | 12 months
  Distance between cementum-enamel junction and gingival margin, measured in millimeters
Bleeding on probing | 12 months
  percentage of sites which bled upon probing

CONTACTS AND LOCATIONS:
Overall Officials: Claudio M Pannuti, PhD, Principal Investigator — University of Sao Paulo; João Batista C Neto, PhD, Study Director — University of Sao Paulo
Locations (1):
- Faculdade de Odontologia da USP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cesar Neto JB, Cavalcanti MC, Silva CO, Almeida VC, Sapata VM, Lazarin RO, Jung R, Romito GA, Tatakis DN, Pannuti CM. Digital three-dimensional assessment of free gingival graft remodeling over 12 months. J Dent. 2024 Sep;148:105216. doi: 10.1016/j.jdent.2024.105216. Epub 2024 Jun 29. PMID 38950768
- [Background] Almeida VC, Pannuti CM, Ferreira MS, Lazarin RO, Romito GA, Jung RE, Tatakis DN, Silva COE, Cesar Neto JB. Conventional versus flap-protected free gingival graft: a multicenter randomized clinical trial. Braz Oral Res. 2023 Jan 6;37:e001. doi: 10.1590/1807-3107bor-2023.vol37.0001. eCollection 2023. PMID 36629587